CLINICAL TRIAL: NCT05344716
Title: Monocentric, Prospective Pilot Study to Test the Efficacy and Safety of the FotonaSmooth Erbium:YAG Laser for the Treatment of Urethral Pain Syndrome in Women
Brief Title: FotonaSmooth Erbium:YAG Laser for the Treatment of Urethral Pain Syndrome in Women
Acronym: UPS-IUL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Prof. Dr. Volker Viereck (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Volker Viereck, Prof. Dr. med., Cantonal Hospital, Frauenfeld
Organization: Cantonal Hospital, Frauenfeld (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pilot UPS-IUL
Record Dates: First submitted 2022-03-30; First posted 2022-04-25 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Pelvic Pain Syndrome
Keywords: urethra; pain; laser; intraurethral; erbium; fotona
MeSH Terms: conditions — Pain | interventions — Lasers

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Laser (Experimental): Intraurethral and vaginal laser treatment
  Interventions: Device: Laser

INTERVENTIONS:
Device: Laser — Intraurethral and vaginal laser treatment

SUMMARY:
Urethral pain syndrome (UPS) is defined by the occurrence of persistent or recurrent episodic urethral pain in the absence of proven infection or other obvious pathology. The objective of this study is to determine the effect of an intraurethral and vaginal laser therapy for the treatment of UPS. The hypothesis is that a significant reduction of urethral pressure pain can be achieved.

DETAILED DESCRIPTION:
Urethral pain syndrome (UPS) is characterized by recurrent or persistent symptoms such as urethral or pelvic pain, daytime frequency and nocturia with unclear aetiology are diagnosed as UPS. Chronic infection by fastidious bacteria leading to chronic inflammation and pain may also cause UPS. Due to the unclear aetiology, the optimal treatment is challenging. It is therefore essential to find new and effective treatment options for patients suffering from UPS. Over the last few years, the use of lasers has become more popular to treat gynaecological and urogynecological conditions including stress urinary incontinence (SUI), genitourinary syndrome of menopause (GSM), vaginal prolapse and other conditions. In several trials, vaginal laser therapy has been shown to have a very good effect on SUI and GSM. Very few publications are available on the use of intraurethral laser therapy for the treatment of SUI and GSM with promising results. This is the first study to test the effect of intraurethral and vaginal laser therapy for the treatment of UPS. The hypothesis is that symptoms can be relieved in patients with UPS i.e. a reduction of urethral pressure pain upon palpation can be achieved.

ELIGIBILITY:
Inclusion Criteria:

* Adult female, 18 years of age or older
* Urethral pressure pain upon palpation, VAS Score ≥ 2
* Intermittent or chronic pain in the urethra and/or the small pelvis (independent of micturition) for at least 6 months
* No significant improvement of UPS from at least one previous conservative treatment (pessary, antibiotics, local oestrogens etc.)
* Signed informed consent

Exclusion Criteria:

* Pregnancy
* Treatment with Isotretinoin (Acne, Rosacea) within last 6 months
* Acute urinary tract infection or other acute infection of the bladder, vagina, vulva or urinary tract detected by routine urine analysis
* Positive urethral swab for Ureaplasma, Mycoplasma or Chlamydia ≤ 6 weeks. Exception: Patients with chronic and persistent fastidious bacteria can be included six weeks after two unsuccessful treatments with antibiotics. Antibiotics therapy must also include sexual partners.
* Pre-existing bladder or urethra pathology
* Interstitial Cystitis
* Endometriosis
* Diagnosis of collagen disorders, e.g. benign joint hypermobility / Elhers-Danlos / Marfans etc.
* Vesicovaginal fistula
* Unwillingness or inability to complete follow-up schedule
* Unwillingness or inability to give informed consent
* Unwillingness or inability to complete questionnaires

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients showing improvement in symptoms due to laser treatment | 5 months
  Reduction of urethral pressure pain upon palpation (visual analogue scale, 0-10 where 0 is none and 10 the worst), cure/improvement defined as >50% reduction compared to baseline

SECONDARY OUTCOMES:
Number of patients showing improvement (reduction) in induration after treatment | 5 months
  digital testing of pelvic induration by physician (scale: high, moderate, none) compared to baseline
Number of patients showing improvement (reduction in questionnaire sum) in symptoms as assed by subjective questionnaire | 5 months, 12 months
  subjective evaluation by validated questionnaire (Genitourinary Pain Index for Women, sum scale 0-45, the lower the value the lower the symptoms) compared to baseline
Number of patients reporting pain during laser treatment | 3 months
  VAS (visual analogue scale, 0-10 where 0 is none and 10 the worst) pain score during laser treatment
Number of patients showing urethral infections before and after treatment | 5 months
  Analysis of urethral infections before and after treatment using urine dipstick test (positive/negative)
Number of patients reporting satisfaction with treatment outcome | 5 months, 12 months
  subjective evaluation of improvement (patient global index fo improvement, 7-item scale from "very much worse" to "very much better"), cure/improvement defined as response "much better" or "very much better"

OTHER OUTCOMES:
Number of patients reprting good tolerability ("good" or "very good") of vulvar creams in combination with laser treatment | 5 months
  Patient satisfaction (5-item scale from "not at all" to "very good") on the use of vulvar creams

CONTACTS AND LOCATIONS:
Overall Officials: Volker Viereck, Prof. Dr., Principal Investigator — Cantonal Hospital, Frauenfeld
Locations (1):
- Cantonal Hospital Frauenfeld, Frauenfeld, Thurgau, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gaspar A, Maestri S, Silva J, Brandi H, Luque D, Koron N, Vizintin Z. Intraurethral Erbium:YAG laser for the management of urinary symptoms of genitourinary syndrome of menopause: A pilot study. Lasers Surg Med. 2018 Oct;50(8):802-807. doi: 10.1002/lsm.22826. Epub 2018 Apr 18. PMID 29667744
- [Background] Gaspar A, Brandi H. Non-ablative erbium YAG laser for the treatment of type III stress urinary incontinence (intrinsic sphincter deficiency). Lasers Med Sci. 2017 Apr;32(3):685-691. doi: 10.1007/s10103-017-2170-5. Epub 2017 Feb 16. PMID 28210823
- [Background] Gaspar A, Silva J, Silva G, Anchelerguez R, Prats J, Sagaz A, Rovere E, Alastra M, Pino J, Jauregui A, Farrugia M, Villaroel F, Guareschi J, Vega M, Biasiori E, Moyano E, La Rosa A, Hreljac I, Vizintin Z. Nonablative transurethral Erbium:YAG laser treatment for chronic prostatitis/chronic pelvic pain syndrome: A prospective comparative study. Neurourol Urodyn. 2021 Jan;40(1):278-285. doi: 10.1002/nau.24551. Epub 2020 Nov 10. PMID 33170523
- [Background] Kuszka A, Gamper M, Walser C, Kociszewski J, Viereck V. Erbium:YAG laser treatment of female stress urinary incontinence: midterm data. Int Urogynecol J. 2020 Sep;31(9):1859-1866. doi: 10.1007/s00192-019-04148-9. Epub 2019 Dec 11. PMID 31828400
- [Background] Yoon SM, Jung JK, Lee SB, Lee T. Treatment of female urethral syndrome refractory to antibiotics. Yonsei Med J. 2002 Oct;43(5):644-51. doi: 10.3349/ymj.2002.43.5.644. PMID 12402379
- [Background] Kaur H, Arunkalaivanan AS. Urethral pain syndrome and its management. Obstet Gynecol Surv. 2007 May;62(5):348-51; quiz 353-4. doi: 10.1097/01.ogx.0000261645.12099.2a. PMID 17425813
- [Background] Gambacciani M, Levancini M. Short-term effect of vaginal erbium laser on the genitourinary syndrome of menopause. Minerva Ginecol. 2015 Apr;67(2):97-102. PMID 25763800
- [Background] Gambacciani M, Levancini M, Cervigni M. Vaginal erbium laser: the second-generation thermotherapy for the genitourinary syndrome of menopause. Climacteric. 2015 Oct;18(5):757-63. doi: 10.3109/13697137.2015.1045485. PMID 26029987
- [Background] Fistonic N, Fistonic I, Gustek SF, Turina IS, Marton I, Vizintin Z, Kazic M, Hreljac I, Perhavec T, Lukac M. Minimally invasive, non-ablative Er:YAG laser treatment of stress urinary incontinence in women--a pilot study. Lasers Med Sci. 2016 May;31(4):635-43. doi: 10.1007/s10103-016-1884-0. Epub 2016 Feb 9. PMID 26861984
- [Background] Fistonic I, Fistonic N. Baseline ICIQ-UI score, body mass index, age, average birth weight, and perineometry duration as promising predictors of the short-term efficacy of Er:YAG laser treatment in stress urinary incontinent women: A prospective cohort study. Lasers Surg Med. 2018 Jan 23. doi: 10.1002/lsm.22789. Online ahead of print. PMID 29360142
- [Background] Gambacciani M, Levancini M, Russo E, Vacca L, Simoncini T, Cervigni M. Long-term effects of vaginal erbium laser in the treatment of genitourinary syndrome of menopause. Climacteric. 2018 Apr;21(2):148-152. doi: 10.1080/13697137.2018.1436538. Epub 2018 Feb 13. PMID 29436235
- [Background] Blaganje M, Scepanovic D, Zgur L, Verdenik I, Pajk F, Lukanovic A. Non-ablative Er:YAG laser therapy effect on stress urinary incontinence related to quality of life and sexual function: A randomized controlled trial. Eur J Obstet Gynecol Reprod Biol. 2018 May;224:153-158. doi: 10.1016/j.ejogrb.2018.03.038. Epub 2018 Mar 22. PMID 29604548